CLINICAL TRIAL: NCT05288062
Title: Evaluating Mechanisms of Immunomodulator Sensitivity and Resistance in Multiple Myeloma
Brief Title: Immunomodulatory Drugs (Lenalidomide With or Without Pomalidomide) in Combination With a Corticosteroid Drug (Dexamethasone) for the Treatment of Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC210809; NCI-2022-01379 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-006597 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-03-03; First posted 2022-03-18 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Plasma Cell Myeloma; Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma; Smoldering Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma | interventions — Biopsy; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (lenalidomide, dexamethasone) (Experimental): Patients with smoldering multiple myeloma receive lenalidomide PO QD alone on days 1-14 OR in combination with dexamethasone PO QD on days 1, 8 and 15. Treatment for cycle 1 continues for 21 days in the absence of disease progression or unacceptable toxicity. Patients then receive lenalidomide PO QD on days 1-21 alone or in combination with dexamethasone PO QD on days 1, 8, 15, and 22, or in combination with another drug. Treatment repeats every 28 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Bone Marrow Biopsy; Drug: Dexamethasone; Drug: Lenalidomide
- Cohort B (lenalidomide, dexamethasone) (Experimental): Patients with newly diagnosed multiple myeloma receive treatment as in Cohort A.
  Interventions: Procedure: Bone Marrow Biopsy; Drug: Dexamethasone; Drug: Lenalidomide
- Cohort C (lenalidomide, dexamethasone, pomalidomide) (Experimental): Patients with relapsed or refractory multiple myeloma receive lenalidomide PO QD on days 1-14 in combination with dexamethasone PO QD on days 1, 8 and 15 OR pomalidomide PO QD on days 1-21 in combination with dexamethasone PO QD on days 1, 8 and 15. Treatment for cycle 1 continues for 21 days in the absence of disease progression or unacceptable toxicity. Patients then receive lenalidomide PO QD on days 1-21 in combination with dexamethasone PO QD on days 1, 8, 15, and 22 OR pomalidomide PO QD on days 1-21 in combination with dexamethasone PO QD on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Bone Marrow Biopsy; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Pomalidomide
- Cohort D (lenalidomide, dexamethasone, pomalidomide) (Experimental): Patients with relapsed multiple myeloma after lenalidomide maintenance receive treatment as in Cohort C.
  Interventions: Procedure: Bone Marrow Biopsy; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Pomalidomide

INTERVENTIONS:
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspirate/biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Dexamethasone — Given orally
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Lenalidomide — Given orally
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Drug: Pomalidomide — Given orally
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst
  Arms: Cohort C (lenalidomide, dexamethasone, pomalidomide); Cohort D (lenalidomide, dexamethasone, pomalidomide)

SUMMARY:
This phase II trial studies the effect of immunomodulatory drug(s) in combination with a corticosteroid drug in treating patients with multiple myeloma or smoldering multiple myeloma. Immunomodulatory drugs such as lenalidomide and pomalidomide work through a variety of mechanisms to affect the function of the immune system. They are widely used as treatment for multiple myeloma and remain the backbone of therapy for both newly diagnosed patients and patients that have multiple myeloma that has come back after treatment (relapsed). Corticosteroid drugs like dexamethasone are strong anti-inflammatory agents that are also widely used to treat patients with multiple myeloma. This study may help doctors find out how patients respond to one treatment cycle of immunomodulatory drug(s) in combination with dexamethasone. This may help doctors determine which combinations of drugs work best in treating patients with multiple myeloma or smoldering multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine response rates (>= partial response [PR]) of prospectively treated multiple myeloma (MM) patients with one cycle of therapy containing a combination of an immunomodulator and dexamethasone.

SECONDARY OBJECTIVE:

I. To identify biomarkers that predict response rates of untreated smoldering MM and MM patients to a combination of an immunomodulator and dexamethasone.

II. To compare response rates of MM among African-Americans (AA) and white patients to a combination of an immunomodulator and dexamethasone.

III. To establish correlation of biomarkers in treated MM patients with the combination of an immunomodulator and dexamethasone to the depth of hematological response observed in new or previously treated patients

OUTLINE: Patients are assigned to 1 of 4 cohorts.

COHORT A: Patients with smoldering multiple myeloma receive lenalidomide orally (PO) once daily (QD) alone on days 1-14 OR in combination with dexamethasone PO QD on days 1, 8 and 15. Treatment for cycle 1 continues for 21 days in the absence of disease progression or unacceptable toxicity. Patients then receive lenalidomide PO QD on days 1-21 alone or in combination with dexamethasone PO QD on days 1, 8, 15, and 22, or in combination with another drug. Treatment repeats every 28 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.

COHORT B: Patients with newly diagnosed multiple myeloma receive treatment as in Cohort A.

COHORT C: Patients with relapsed or refractory multiple myeloma receive lenalidomide PO QD on days 1-14 in combination with dexamethasone PO QD on days 1, 8 and 15 OR pomalidomide PO QD on days 1-21 in combination with dexamethasone PO QD on days 1, 8 and 15. Treatment for cycle 1 continues for 21 days in the absence of disease progression or unacceptable toxicity. Patients then receive lenalidomide PO QD on days 1-21 in combination with dexamethasone PO QD on days 1, 8, 15, and 22 OR pomalidomide PO QD on days 1-21 in combination with dexamethasone PO QD on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.

COHORT D: Patients with relapsed multiple myeloma after lenalidomide maintenance receive treatment as in Cohort C.

After completion of study treatment, patients are followed up within 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* COHORT A: Patient must have untreated smoldering multiple myeloma which is defined by the presence of 10% or more but less than 60% clonal plasma cells in the bone marrow and the absence of any of the following myeloma related symptoms or laboratory and radiographic abnormalities: anemia, hypercalcemia, renal insufficiency, hypercalcemia, serum free light chain ratio of greater than 100 or more than one focal marrow multiple myeloma lesion on magnetic resonance imaging (MRI)
* COHORT B: Patient must have newly diagnosed myeloma requiring treatment and no prior therapies
* COHORT C: Patient must have relapsed or refractory multiple myeloma with at least one prior therapy for their multiple myeloma but not refractory to all IMiDs
* COHORT D: Patient must have relapsed or refractory multiple myeloma with lenalidomide as part of a maintenance regimen as their most recent therapy
* Measurable disease
* Provide written informed consent
* Patient must be considered for treatment with an IMiD containing regimen
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, 2 or 3
* Hemoglobin >= 9.0 g/dL (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless due to Gilbert's syndrome, in which case the direct bilirubin must be =< 1.5 X ULN (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) 3 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =< 14 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy (obtained =< 14 days prior to registration)
* Calculated creatinine clearance >= 45 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willingness to provide mandatory blood and bone marrow specimens for correlative research
* Willing to follow the requirements of the Pomalyst Risk Evaluation and Mitigation Strategy (REMS) program

Exclusion Criteria:

* An agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* History of myocardial infarction =< 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilson I. Gonsalves, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (4):
- United States (4):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A (Lenalidomide, Dexamethasone) | Cohort B (Lenalidomide, Dexamethasone) | Cohort C (Lenalidomide, Dexamethasone, Pomalidomide) | Cohort D (Lenalidomide, Dexamethasone, Pomalidomide)
Started | 0 | 5 | 12 | 0
Completed | 0 | 5 | 10 | 0
Not Completed | 0 | 0 | 2 | 0
Not completed — Ineligible | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only patients that completed the study were included in analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Lenalidomide, Dexamethasone) | Cohort B (Lenalidomide, Dexamethasone) | Cohort C (Lenalidomide, Dexamethasone, Pomalidomide) | Cohort D (Lenalidomide, Dexamethasone, Pomalidomide) | Total
Number analyzed (Participants) | 0 | 5 | 10 | 0 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 61.4 (15.2) | 69.9 (12.1) |  | 67.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 0 | 5
  Male | 0 | 3 | 7 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 1 | 1 |  | 2
  Not Hispanic or Latino |  | 4 | 9 |  | 13
  Unknown or Not Reported |  | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 |  | 0
  Asian |  | 1 | 0 |  | 1
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 |  | 0
  Black or African American |  | 0 | 1 |  | 1
  White |  | 3 | 9 |  | 12
  More than one race |  | 0 | 0 |  | 0
  Unknown or Not Reported |  | 1 | 0 |  | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 5 | 10 |  | 15

OUTCOME MEASURES:

1. Primary Outcome: Response Rates (RR) at First Assessment
Description: RR is defined as a binary variable. A success will be defined as patient who achieve a response of a partial response (PR) or better using the International Myeloma Working Group (IMWG) criteria. Biomarkers of interest will be identified and categorized into clinically relevant groups (e.g. positive vs. negative) by evaluating baseline and post treatment (after cycle one) biospecimens. RR will be estimated within each biomarker. Each cohort (A-D) will be evaluated separately and independently.
Time Frame: 21 days
Population: Only patients that completed the study were included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Lenalidomide, Dexamethasone) | Cohort B (Lenalidomide, Dexamethasone) | Cohort C (Lenalidomide, Dexamethasone, Pomalidomide) | Cohort D (Lenalidomide, Dexamethasone, Pomalidomide)
Number analyzed (Participants) | 0 | 5 | 10 | 0
Participants |  | 1 | 4 |

2. Secondary Outcome: Predictive Biomarkers
Description: Biomarkers and RR will be analyzed using logistic regressions to identify predictive biomarkers.
Time Frame: Up to 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Response Rates (RR) Among African American (AA) and White Patients
Description: Chi-square (or Fischer Exact) test and 95% confidence intervals will be estimated to compared AA and white patients descriptively.
Time Frame: Up to completion of 1 cycle of treatment (21 days)
Reporting Status: Not Posted

4. Secondary Outcome: Depth of Hematological Responses
Description: Correlation between the depth of hematological responses and biomarkers will be estimated. Logistic regressions and chi square (or Fischer exact) testing will be utilized.
Time Frame: Up to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Cohort B (Lenalidomide, Dexamethasone): Patients with newly diagnosed multiple myeloma receive treatment as in Cohort A.
  Bone Marrow Biopsy: Undergo bone marrow aspirate/biopsy Dexamethasone: Given orally Lenalidomide: Given orally
- Cohort C (Lenalidomide, Dexamethasone, Pomalidomide): Patients with relapsed or refractory multiple myeloma receive lenalidomide PO QD on days 1-14 in combination with dexamethasone PO QD on days 1, 8 and 15 OR pomalidomide PO QD on days 1-21 in combination with dexamethasone PO QD on days 1, 8 and 15. Treatment for cycle 1 continues for 21 days in the absence of disease progression or unacceptable toxicity. Patients then receive lenalidomide PO QD on days 1-21 in combination with dexamethasone PO QD on days 1, 8, 15, and 22 OR pomalidomide PO QD on days 1-21 in combination with dexamethasone PO QD on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity.
  Bone Marrow Biopsy: Undergo bone marrow aspirate/biopsy Dexamethasone: Given orally Lenalidomide: Given orally Pomalidomide: Given orally
Arm/Group | Cohort B (Lenalidomide, Dexamethasone) | Cohort C (Lenalidomide, Dexamethasone, Pomalidomide)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/5 | 2/11
Other Adverse Events (participants affected / at risk) | 3/5 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort B (Lenalidomide, Dexamethasone) (N=5) | Cohort C (Lenalidomide, Dexamethasone, Pomalidomide) (N=11)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort B (Lenalidomide, Dexamethasone) (N=5) | Cohort C (Lenalidomide, Dexamethasone, Pomalidomide) (N=11)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 4 (4)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (2)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 3 (4)
Neutrophil count decreased (Investigations) | 1 (1) | 4 (7)
White blood cell decreased (Investigations) | 2 (2) | 2 (5)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT05288062/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT05288062/ICF_001.pdf